CLINICAL TRIAL: NCT04730063
Title: Prospective Non-Interventional Study Evaluating Non-invasive Measurements of Pulmonary Blood Flow, Functional Residual Capacity, Shunt Fraction Index and Airway Dead Space Measured With the VQm PHM™ to Clinical Gold Standards
Brief Title: Evaluation of Novel Cardio-Pulmonary Physiological Monitor, the VQm PHM™, for Acute Care Medicine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rostrum Medical Innovations Inc. (Industry)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1685958-2
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Elective Procedures Requiring Mechanical Ventilation
Keywords: Physiologic Monitors; Acute Care Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: VQm PHM™ — Procedure: Non-invasive measurements obtained with the VQm PHM™

SUMMARY:
This is a prospective, observational study to assess agreement of pulmonary health parameters measured by a new non-invasive physiologic monitor, the VQm pulmonary health monitor (PHM)™ with clinical gold standards.

DETAILED DESCRIPTION:
The specific aim of this study is to evaluate the intermittent non-invasive measurements of pulmonary function: pulmonary blood flow (PBF), functional residual capacity (FRC), shunt fraction index (Qsi) and airway dead space measured by the VQm PHM™ compared to known clinical standards. PBF will be compared to continuous and intermittent bolus thermodilution cardiac output as measured through a Swan-Ganz catheter. FRC will be compared to an FRC measurement provided by a standard nitrogen washout method. Qsi will be compared to shunt fraction calculated through mixed venous and arterial blood gas values (VBGs/ABGs). Airway dead space will be compared to an airway dead space measurement provided by a ventilator.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Scheduled for an elective surgical procedure with an anticipated duration of more than 2 hours requiring general anesthesia without the use of inhalation anesthetics
* Surgical procedure that requires pressure-controlled positive pressure ventilation using an endotracheal tube
* Surgical procedure that requires the use of intra-arterial pressure monitoring and/or a Swan-Ganz catheter for the monitoring of continuous cardiac output

Exclusion Criteria:

* Patients who require ventilation tidal volumes less than 250cc
* Age less than 18 years
* Pregnancy
* Prisoners
* Surgical procedure which requires carbon dioxide (CO2) insufflation
* Unable to tolerate a transient increase in inhaled CO2
* Unable to tolerate a transient increase in inhaled nitrous oxide (N2O) or use of N2O is contraindicated
* Patients who require a high fraction of inspired oxygen (FiO2) (>70%) to maintain a hemoglobin saturation (SpO2>98%)

Women, minorities or non-English speaking subjects will not be excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery requiring mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of pulmonary function parameters to known clinical standards | Through study completion, an average of 12 months
  Assess agreement between measurements from VQm PHM™ to clinical gold standards

CONTACTS AND LOCATIONS:
Overall Officials: Neal W Fleming, M.D., Ph.D., Principal Investigator — Director, Cardiovascular and Thoracic Anesthesiology
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States